CLINICAL TRIAL: NCT05543824
Title: Hemodynamic Impact of Epidural Anesthesia in Relation to Age in Pediatric Patients.
Acronym: REHAEPP-2022
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Daniel Pérez, M.D., Hospital Universitario La Fe
Other Study IDs: REHAEPP-2022
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Hemodynamic Monitoring; Anesthesia; Adverse Effect; Pediatric Major Surgery; Epidural Analgesia
Keywords: Pediatric surgery; Epidural analgesia; Hemodynamic monitoring
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Epidural and arterial catheter: Patients who require placement of an epidural catheter to control postoperative pain and invasive blood pressure will be identified, allowing advanced monitoring using the MostCare Up® device. After identification, the objective of the study will be explained and their consent will be requested to collect the data after the intervention, recording the hemodynamic data before and after the initial bolus of local anesthetic administered: 0.25% levobupivacaine, the dose of which is calculated with the Takasaki formula: 0.05ml x weight (kg) x number of dermatomes to anesthetize.
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — Patients who require placement of an epidural catheter to control postoperative pain and invasive blood pressure will be identified, allowing advanced monitoring using the MostCare Up® device. After identification, the objective of the study will be explained and their consent will be requested to collect the data after the intervention, recording the hemodynamic data before and after the initial bolus of local anesthetic administered: 0.25% levobupivacaine, the dose of which is calculated with the Takasaki formula: 0.05ml x weight (kg) x number of dermatomes to anesthetize
  Other Names: epidural catheter; invasive arterial catheter

SUMMARY:
Epidural analgesia is established as the gold standard in the management of post-surgical pain in multiple modalities, including the pediatric patient. It is a technique that is not without risks, but with multiple benefits such as less response to stress, less incidence of chronic pain after surgery, less incidence of nausea and vomiting and other adverse effects derived from opioids, faster recovery and increased patient and family satisfaction.

However, as it has been mentioned, the epidural carries risks both in the technique itself (wet or intravascular puncture) and subsequently after the injection of medication that generates a sympathetic blockade with arterial hypotension and an increase in compensatory heart rate. Unlike in adult patients, in pediatric patients epidural and subarachnoid anesthesia are better tolerated hemodynamically due to less vagal and sympathetic activity and almost no systemic venodilation. This lower activity of the autonomic nervous system is due to its immaturity, which is why, with the growth of the infant, this anesthetic technique increasingly affects its hemodynamics, being similar to the adult at the age of 8-12 years.

The study hypothesis does not differ from that stated in physiology books and studies, but the investigators seek to identify the direct correlation of age with the different hemodynamic parameters available with current technology (cardiac output, systemic vascular resistance, blood pressure ) in pediatric patients after epidural anesthesia.

The study will be carried out in pediatric patients undergoing major surgery that requires the placement of an epidural catheter and invasive blood pressure, without modifying in any way the usual practice of the responsible anesthesiologist. The patient's hemodynamic data will be collected at time 0 (prior to catheter placement), one minute, 5 and 10 minutes after the bolus of local anesthetic administered to measure the child's hemodynamic response and relate it to their age and development. .

DETAILED DESCRIPTION:
Through this work the investigators seek to establish statistically and numerically a hypothesis affirmed in physiology books. In this way, if it is found a positive correlation with age and hypotension, the responsible physician can be alerted to the need for possible vasoconstrictor requirements or more advanced monitoring in order to reduce intraoperative risks.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 12 years of age undergoing major surgery with epidural catheter placement and invasive blood pressure.

Exclusion Criteria:

* Allergy to local anesthetics (LA).
* Congenital diseases which affect the central nervous system.
* Inability to place an invasive arterial catheter.

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients under 12 years of age undergoing major surgery in the University Hospital La Fe, in Valencia
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-04-18 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic repercussion | time zero until 10 minutes
  Drop in blood pressure after epidural levobupivacaine bolus
Age related repercussion | 0 years until 12 years
  Relate the blood pressure drop to the age of the patient

SECONDARY OUTCOMES:
Epidural level | time zero until 10 minutes
  Asses if the epidural level (lumbar or thoracic) influence the different results
Gender | time zero until 10 minutes
  Asses if the gender of the patient influence the different results

CONTACTS AND LOCATIONS:
Locations (1):
- Daniel Perez Ajami, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gootman PM, Gootman N, Buckley BJ. Maturation of central autonomic control of the circulation. Fed Proc. 1983 Apr;42(6):1648-55. PMID 6832381
- [Background] Martinez-Telleria A., Cano Serrano M.E.: Anestesia epidural lumbar. En Anestesia Locorregional en Pediatria, Blanco Vargas D., Reinoso Barbero F., Cruz Tejado J. Ed. ARAN, 2005, Madrid, Cap.9: 129-143.
- [Background] Alonso-Inigo JM, Escriba FJ, Carrasco JI, Fas MJ, Argente P, Galvis JM, Llopis JE. Measuring cardiac output in children undergoing cardiac catheterization: comparison between the Fick method and PRAM (pressure recording analytical method). Paediatr Anaesth. 2016 Nov;26(11):1097-1105. doi: 10.1111/pan.12997. Epub 2016 Aug 27. PMID 27565740